CLINICAL TRIAL: NCT02883101
Title: The Effects of Pulmonary Rehabilitation in Patients With Non-cystic Fibrosis Bronchiectasis: A Randomised Controlled Trial
Brief Title: The Effects of Pulmonary Rehabilitation in Patients With Non-cystic Fibrosis Bronchiectasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: All India Institute of Medical Sciences (Other)
Responsible Party: Principal Investigator, Dr. Rohit Kumar, Senior Resident, All India Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IESC/T-345
Record Dates: First submitted 2016-08-14; First posted 2016-08-30 (Estimated); Last update posted 2017-07-05 (Actual); Status verified 2017-07

CONDITIONS: Non-cystic Fibrosis Bronchiectasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pulmonary rehabilitation group (Active Comparator): Participants randomised to the PR group will receive exercise training and regular instruction in self-management of ACT along with standard care. Patients will be enrolled into the pulmonary rehabilitation programme, in the Department of Pulmonary Medicine and Sleep disorders, All India Institute of Medical Sciences.
  The total duration of the programme would be 8 weeks, with thrice weekly sessions of exercise training of 1 hour duration each. Of these sessions, at least 2 will be supervised while one will be at home. The patient will be asked to maintain a personal log recording the date, time, duration and type of exercise performed to ensure compliance, and these will be regularly reviewed and monitored.
  The Rehabilitation Programme will include the following:
  i. Patient education ii. Exercise training iii. Ventilator and breathing exercises
  Interventions: Behavioral: Pulmonary Rehabilitation
- Standard care group (No Intervention): Candidates randomized to the "standard care group" will receive standard care for bronchiectasis according to current guidelines. These participants will receive instruction and review of airway clearance therapy (ACT). Each participant will be provided with written information about bronchiectasis and education regarding self-management of the condition. Participants who have not been previously instructed in any ACT will be taught the active cycle of breathing technique. These participants will not receive any supervised exercise training.

INTERVENTIONS:
Behavioral: Pulmonary Rehabilitation — The Rehabilitation Programme will include the following :
  i. Patient education ii. Exercise training iii. Ventilator and breathing exercises
  Other Names: The Rehabilitation Programme
  Arms: Pulmonary rehabilitation group

SUMMARY:
Number of Patients:

Study group - Bronchiectasis that is not attributable to Cystic fibrosis

* Group 1 - Pulmonary Rehabilitation
* Group 2 - Standard care

Sample size - 20 in each arm

Study Design:

* Randomised controlled trial (RCT)

All patients who qualify for the study will undergo a detailed evaluation. Baseline assessment will include the following parameters:

* Anthropometry
* Pulmonary Function Tests and Respiratory muscle strength
* Cardiopulmonary Exercise Testing (CPET)
* Six Minute Walk Test (6MWT)
* Severity of dyspnoea (Dyspnoea scale)
* Limb muscle strength
* Inflammatory markers in the serum - C-reactive protein
* Quality of Life

Patients will then be randomized (using table of random numbers) to either the pulmonary rehabilitation group or the standard arm group. After 8 weeks of pulmonary rehabilitation, patients will again be reassessed by the aforementioned tools.

DETAILED DESCRIPTION:
METHODOLOGY

Type of study - Randomised controlled trial (RCT)

Study period - March 2014 to July 2016

Place of study - Department of Pulmonary Medicine and Sleep Disorders, All India Institute of Medical Sciences, New Delhi

Study group - Bronchiectasis that is not attributable to Cystic fibrosis

* Group 1 - Pulmonary Rehabilitation (PR)
* Group 2 - Standard care

Sample size - 20 in each arm

The study requires patients to attend the pulmonary rehabilitation program twice a week for 8 weeks.

Consent will be taken from all patients prior to enrollment.

Exacerbations of bronchiectasis will be defined by the following criteria:

At least four of the following clinical signs and symptoms suggestive of an acute exacerbation of bronchiectasis over two consecutive days:

* Increase in sputum quantity
* Change in sputum colour
* Change in sputum viscosity
* Increase in cough
* Increase in dyspnoea
* Increase in fatigue/lethargy
* Fever (self-reported)
* Episode of haemoptysis

The number of acute pulmonary exacerbations per year in the previous years will be recorded.

All patients attending the out patient department of pulmonary department of All India Institute of Medical Sciences will be screened for recruitment in the study.

Baseline evaluation

All patients who qualify for the study will undergo a detailed evaluation. This will include demographic data, complete medical history and clinical examination including anthropometry. Baseline assessment will include the following parameters:

i. Anthropometry

ii. Pulmonary Function Tests and Respiratory muscle strength

iii. Cardiopulmonary Exercise Testing (CPET)

iv. Six Minute Walk Test (6MWT)

v. Severity of dyspnoea (Dyspnoea scale)

vi. Limb muscle strength

vii. Inflammatory markers in the serum - C-reactive protein

viii. Quality of Life

The participants will then be randomly assigned to receive either standard care alone or pulmonary rehabilitation. The randomisation will be completed by the creation of a random numbers table.

Intervention

Standard care group

Candidates randomized to the "standard care group" will receive standard care for bronchiectasis according to current guidelines. These participants will receive instruction and review of airway clearance therapy (ACT). Each participant will be provided with written information about bronchiectasis and education regarding self-management of the condition. Participants who have not been previously instructed in any ACT will be taught the active cycle of breathing technique. These participants will not receive any supervised exercise training.

Pulmonary rehabilitation group

Participants randomised to the Pulmonary Rehabilitation group will receive exercise training and regular instruction in self-management of ACT along with standard care. Patients will be enrolled into the pulmonary rehabilitation programme, in the Department of Pulmonary Medicine and Sleep disorders, All India Institute of Medical Sciences.

The total duration of the programme would be 8 weeks, with thrice weekly sessions of exercise training of 1 hour duration each. Of these sessions, at least 2 will be supervised while one will be at home. The patient will be asked to maintain a personal log recording the date, time, duration and type of exercise performed to ensure compliance, and these will be regularly reviewed and monitored.

The Rehabilitation Programme will include the following:

i. Patient education

ii. Exercise training

iii. Ventilator and breathing exercises

Outcome Assessment

The patients will be reassessed at the end of the 8 week training programme.

Primary outcome measures:

* Maximum exercise capacity - measured with the 6MWT (the primary outcome is the greatest distance walked) and the CPET (VO2 max)
* HRQoL measured with the St. George Respiratory Questionnaire

Secondary outcome measures:

* Change in the Leicester Cough Questionnaire
* Change in the C- reactive protein
* Change in the lung Functions
* Change in the anxiety and depressions score
* Change in the hand grip dynamometry

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Diagnosed bronchiectasis that is not attributable to cystic fibrosis, confirmed radiologically on high resolution computed tomography
* Exertional dyspnoea (Modified Medical Research Council (mMRC) score ≥ 2 and a history of at least two exacerbations in the past year
* Willing to give informed consent

Exclusion Criteria:

* Smoking history ≥ 10 pack years or physician diagnosis of chronic obstructive pulmonary disease
* A clinical diagnosis of asthma
* Interstitial lung disease (clinical/radiological diagnosis)
* Medical conditions which could place the individual at risk during exercise testing or training (eg. angina) or conditions that may restrict the participant's ability to exercise (eg. severe orthopaedic or neurologic impairments);
* Participation in a PR program within the last 12 months.
* Patient having an exacerbation of bronchiectasis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-06; Primary Completion 2016-10 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Exercise capacity | 8 weeks
  Assessed using 6 minute walk distance and cardiopulmonary exercise testing

SECONDARY OUTCOMES:
Cough related QoL | 8 weeks
  Assessed using Leicester Cough Questionnaire
Health Related Quality of Life | 8 weeks
  Assessed using St George Respiratory questionnaire
Lung Functions | 8 weeks
  Assessed using pulmonary function testing
Anxiety and depressions score | 8 weeks
  Assessed using Depression Anxiety and Stress Scale (DASS)

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Rohit Kumar, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: No